CLINICAL TRIAL: NCT02313805
Title: The Effect of a Checklist on the Quality of Education During Insulin Initiation by Trained Medical Students: a Randomized Controlled Trial
Brief Title: The Effect of a Checklist on the Quality of Education During Insulin Initiation by Trained Medical Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: UndergradStudy
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus
Keywords: Insulin initiation; Insulin checklist
MeSH Terms: conditions — Diabetes Mellitus | interventions — Checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With checklist (Experimental): Students will simulate insulin initiation with the aid of a checklist
  Interventions: Other: Checklist
- Without checklist (No Intervention): Students will simulate insulin initiation without the aid of a checklist

INTERVENTIONS:
Other: Checklist — The checklist is a simple A4 size, two sided, document. Eleven checklist items covering twenty-one key educational points are on the front. Images illustrating the process of using a syringe to draw up insulin from a vial as well as injection sites (for children, adults and pregnant women) are on the back.
  Other Names: Insulin initiation checklist
  Arms: With checklist

SUMMARY:
Diabetes prevalence continues to rise worldwide, leading to the increasing use of insulin. This especially applies to developing countries where the needle-and-syringe method of administration remains the most affordable and effective form of hyperglycemic treatment. Competent health care professionals are required to ensure safe insulin initiation. The investigators will evaluate a teaching intervention on insulin initiation for medical students, and whether after experiencing that intervention the use of a checklist, during simulate insulin initiation, improves the education they provide to patients.

DETAILED DESCRIPTION:
Introduction:

Diabetes is on the increase worldwide. The International Diabetes Federation estimates that there are currently 382 million persons diagnosed with diabetes. The prevalence is expected to increase to over 592 million in less than 25 years [1]. This increase is disproportional in the developing world, with 80% of those affected living in low- and middle-income countries. For example, in South and Central America, the prevalence of diabetes is estimated to increase by over 60% in the next two decades [2].

Insulin is one of the agents that can be used in the treatment of diabetes mellitus. Diabetes is characterized by a progressive decline in beta-cell function and insulin secretion. Over time, a significant number of persons with diabetes will require intensification of management, and possibly insulin treatment to achieve acceptable glycemic control [3]. Insulin remains the oldest and most effective treatment of hyperglycemia. It is also possibly the cheapest form of treatment relative to its potency, particularly when used in its animal or human forms.

Insulin is a particularly important treatment option in the developing world and in low-income groups in the developed world. In the developing world, drug affordability has limited the international evolution from an algorithmic to an individualized approach to glycemic management [4, 5]. In many countries, insulin remains the affordable second or third line choice for treatment, and will therefore be used with greater frequency.

Insulin initiation is, however, a complex task. To safely initiate insulin, many important aspects of patient education must be addressed. Patients must understand the technicalities of drawing insulin with a needle and syringe as well as administering insulin with a syringe, pen or pump. The side effects of weight gain and hypoglycemia must also be understood, including the recognition and treatment of the latter.

Checklists have been shown to increase the quality of care by reducing errors [6]. They reduce the cognitive load of decision making by decreasing analytic conscious thinking [7]. At the most basic level, they can reduce human error by providing a documented methodological approach to completing tasks. This advantage may be useful in the complex and potentially dangerous arena of insulin initiation.

We seek to evaluate a teaching intervention on insulin initiation, and to determine whether there are safety gains to the additional use of a checklist. This evaluation will be done by means of patient simulations, which allow reliable evaluation [8] without exposing patients to risks [9].

Research hypothesis (alternate):

Using a checklist during insulin initiation, with a needle and syringe, can improve patient education on safe and effective insulin use, above that of thorough undergraduate education.

Methods:

Trial design; The study is randomized and controlled. Initially, the students will all experience a two-hour training session on insulin initiation. Within a week of completing the training, they will be asked to submit a 250 to 400-word reflective narrative, with guiding questions for reflection.

Two to four weeks after training, students consenting to participate in the study will be randomly assigned to the two study groups: the control group and the intervention group. They will be asked to complete a simulation exercise on insulin initiation, with (intervention group) or without (the control group) the availability of an insulin initiation checklist. Performance during each simulation will be assessed with the aid of a check sheet.

The Checklist; The checklist was developed by a task-force, which consisted of eleven individuals: a layperson, a pharmacist, two dietitians, two diabetes educators, a podiatrist, a diabetes specialist nurse, a pediatrician and two diabetologists. The process was lead by the pharmacist, diabetes specialist nurse and one of the diabetologists. The final version of the checklist was achieved through iterative cycles of re-design and feedback. The aim was to develop a simple A4-size, two-sided document that could be easily copied. Eleven checklist items were agreed upon, which cover insulin side effects; use and disposal of syringes; insulin administration and storage; and the recognition and treatment of hypoglycemia. Images illustrating the process of using a syringe to draw insulin from a vial as well as injections sites (for children, adults and pregnant women) were included at the back. There was also space provided for documentation of the client's name and registration number, insulin type and when it should be taken, medications to be stopped, and the date and signature of the facilitator.

The Check Sheet; A check sheet will be used to evaluate the performance of the undergraduate students during each simulation. Educational tasks will be listed under five sub-headings: 'side effects', 'hypoglycemia', 'drawing up insulin', 'insulin administration', and 'other'. Tick boxes will be used to 'check off' whether tasks are performed adequately, inadequately or not at all. Each task will have brief notes on what constitutes adequate performance.

Setting and Simulation; The study will take place within a nine-week final year medicine clerkship at the University of the West Indies, Cave Hill, Barbados. Every nine weeks, the simulation will take place within the medicine end-of-clerkship Objective Structured Clinical Examination. An actor/actress will be used during the simulations to play the role of the patient, in which he/she will require education on the use and administration of insulin via a needle and syringe. The participant will be given instructions for the simulation and the use of the checklist, if in the intervention group.

Training session on insulin initiation; Key aspects of the lesson plan will be as outlined below:

Time: 120 minutes Number of students: 7 to 10

Materials:

* Insulin bottles
* At least 7 insulin syringes
* An orange or suitable model for injecting
* 7 to 10 insulin initiation checklists
* 7 to 10 instruction sheets for the simulation of section F
* Sharps disposal container

Aim: To be able to competently initiate insulin in clients with diabetes

Outcomes: Ability to,

1. Evaluate clients to determine whether insulin initiation is appropriate
2. Evaluate clients and decide on how insulin will be initiated and titrated
3. Discuss the major side effects of insulin use, including weight gain and hypoglycemia
4. Discuss the frequency and timing of glucose monitoring on insulin regimes (background, biphasic and basal bolus)
5. Explain to clients how to recognize and treat hypoglycemia
6. Demonstrate and explain to clients the proper technique of drawing up and injecting insulin, using a needle and syringe as well as pen

Learning methods:

* Case based approach
* Socratic discussion
* Use of simulation to create a clinically authentic learning environment
* Kolb's experiential reflective cycle
* Utilization of checklist to structure learning

Session structure:

A: (10 minutes) Brief review of insulin types

B: (30 minutes - 10 minutes per case)

Discussion of three clinical case scenarios, to decide on:

1. whether insulin initiation is appropriate and which regime should be used,
2. the frequency of glucose monitoring and,
3. the approach to initiation and titration of insulin, if applicable

General learning points from this section

Indications of insulin:

* Type-1 diabetes
* Diabetes due to pancreatic insufficiency
* Type-2 diabetes not adequately controlled on oral agents (as second-line or third-line agent) when insulin can be safely introduced

Weight gain with insulin is approximately 2 to 4 kg and proportional to glucose lowering. It is likely due to reduction in glycosuria.

C: (15 minutes) Students are to discuss key elements of education for a client who is learning to draw and self-administer insulin, using a needle and syringe.

D: (10 minutes) Simulation- students are to demonstrate how they would educate a client who is to be started on insulin using needle and syringe. Instructions given to students: please start this patient on 10 units of Novolin N at bedtime; administration will be by the needle and syringe method; and, please provide any education required. A diabetes specialist nurse (DSN) will act as the simulated client. Other students will observe and reflect on how they would do it.

E: (30 minutes) Insulin initiation will be taught by DSN, using the structure of the checklist. Methods of administration will include syringe and pen.

F: (30 minutes - Role change at 15 minutes) Simulation- Students are to work in pairs, one acting as the patient and one the doctor, to simulate the education required during insulin initiation. "Doctors" are to have instructions and to use the checklist during the process of initiation.

Insulin initiation reflective narrative:

Instructions to students; Having experienced the insulin initiation session you are now required to write a short, 250-400 word reflective narrative. The desired outcome of this process is enhancement of your understanding of what you learnt, what further knowledge and skills are needed and what facilitated your learning. Please consider the guiding questions below to assist this process.

1. How did the session impact my knowledge or skills of insulin initiation?
2. What further actions will enable me to provide the best quality care during insulin initiation?
3. What made the session a useful learning experience for me?

Please note that the submission of an adequate piece is an essential part of the educational intervention and this will be assessed on the presence of content related to the above questions.

Evaluation:

The educational intervention will be evaluated on 2 of the 4 levels of the Kirkpatrick evaluation model 10. On level one, content analysis of the reflective narrative will provide information on what was liked about the intervention. On level two, student's performance during simulation of insulin initiation will provide information on what was learnt. Additionally, comparison of the students initiating insulin with and without (the control group) a checklist will give insight on safety gains with its use.

Analysis:

Reflective commentaries will be analyzed qualitatively using Atlas ti V7 software. Code list creation will be both inductive (codes formulated based on the research question and available literature) and deductive (codes based on other information derived from the commentaries). Thematic analysis will take place through iterative cycles of coding, updating of codes and analysis. To ensure consistency in the analytic process, two researchers will participate in this process and meet regularly to compare analyses within and across participants. A third researcher will repeat the analysis in the event of discrepancies.

Quantitative data will be analyzed using SPSS version 18 (IBM Inc., Armonk, New York, USA). Descriptive statistics will be used to describe performance without the checklist. The chi-squared test will be used to analyze nominal data captured with and without the use of the checklist. If the necessary assumptions apply the t-tests will determine whether there are statistically significant differences within checklist scores between the administrations in each group. If the necessary assumptions do not apply the Wilcoxon signed-rank test will be used respectively. A p-value of < 0.05 will be considered to represent statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students in their final-year medicine clerkship at the University of the West Indies, who are within one year of starting supervised post-graduate employment (internship).
* Students who consent to participate in the study (voluntary participation only).

Exclusion Criteria:

* Students who refuse consent to participate in the study.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The total number of educational points addressed for the safe and effective use of insulin (of the possible 21 specified) | 2 years

SECONDARY OUTCOMES:
The number of educational points addressed under each of the four educational domains: insulin side effects, recognition and treatment of hypoglycemia, administration of insulin, and drawing up insulin using the syringe method. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles G Taylor Jr, MBBS MA MRCP, Principal Investigator — University of the West Indies, Cave Hill
Locations (1):
- The University of the West Indies, Cave Hill Campus, Bridgetown, Saint Michael, Barbados

REFERENCES:
- [Background] 1. International Diabetes Federation. IDF Diabetes Atlas 6th Edition <http://www.idf.org/diabetesatlas>. Accessed May. 2013.
- [Background] 2. [Anonymous]IDF Diabetes Atlas. Fifth Edition ed. 2011.
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Qaseem A, Humphrey LL, Sweet DE, Starkey M, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Oral pharmacologic treatment of type 2 diabetes mellitus: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2012 Feb 7;156(3):218-31. doi: 10.7326/0003-4819-156-3-201202070-00011. PMID 22312141
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] 6. Gawande A. The Checklist Manifesto: How to Get Things Right. NY: Metropolitan Books, 2009.
- [Background] Ely JW, Graber ML, Croskerry P. Checklists to reduce diagnostic errors. Acad Med. 2011 Mar;86(3):307-13. doi: 10.1097/ACM.0b013e31820824cd. PMID 21248608
- [Background] 8. Harden, J.,P.Collins, R.M. AMEE medical education guide no. 13: Real patients, simulated patients and simulators in clinical examinations. Med Teach. 1998; 20:508-521.
- [Background] Cleland JA, Abe K, Rethans JJ. The use of simulated patients in medical education: AMEE Guide No 42. Med Teach. 2009 Jun;31(6):477-86. doi: 10.1080/01421590903002821. PMID 19811162
- [Background] 10. Kirkpatrick DL, Kirkpatrick JD. Implementing the Four Levels: A Practical Guide for Effective Evaluation of Training Programs. 235 Montgomery Street, Suite 650, San Francisco, CA 94104-2916: Berrett-Koehler Publishers, Inc., 2007.